CLINICAL TRIAL: NCT00391547
Title: Phase II Pilot Efficacy Study to Treat Gingivitis
Brief Title: Pilot Efficacy Study to Treat Gingivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biomedical Development Corporation (Industry)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 0609059R44NR009015-02; NIH Grant No. 9R44NR009015-02
Record Dates: First submitted 2006-10-20; First posted 2006-10-24 (Estimated); Last update posted 2007-10-22 (Estimated); Status verified 2007-10

CONDITIONS: Gingival Diseases
Keywords: Gingivitis Disease
MeSH Terms: conditions — Gingival Diseases

INTERVENTIONS:
Drug: Frio Oral Rinse

SUMMARY:
The primary purpose is to demonstrate the efficacy of a prescription mouthrinse in human subjects for treatment of Gingivitis.

DETAILED DESCRIPTION:
Gingivitis is an endemic disease that is a precursor to periodontal disease. Two mouthrinse agents, Peridex and Listerine, have received the Seal of Acceptance from the Council on Dental Therapeutics of the American Dental Association for the control of supragingival plaque and gingivitis. Peridex (0.12% chlorhexidine, bisbiguanide cationic detergent) is a prescription mouthrinse that demonstrates potent anti-plaque and anti-gingivitis action. Chlorhexidine rinses are also prescribed to prevent post surgical infections. Chlorhexidine has broad spectrum antibacterial activity and substantivity. With prolonged use, chlorhexidine maintains its effectiveness but causes staining of natural teeth and composite materials used in restorative dentistry. Other side effects associated with chlorhexidine are calculus formation and possible alterations in taste. Although chlorhexidine rinses and supragingival irrigations have demonstrated significant efficacy in reducing plaque and gingivitis, chlorhexidine has had a minimal impact in treating periodontal disease. Listerine, comprised of essential oils, is an over-the-counter mouthrinse that is less effective than chlorhexidine in controlling plaque and gingivitis, but has minimal side effects. Other agents such as quaternary ammonium compounds and metal salts are rarely used alone but can be used in combination with other antimicrobial rinses to enhance their effectiveness.

ELIGIBILITY:
Inclusion Criteria:

Subjects shall meet all of the following inclusion criteria to be eligible for participation in this study:

* Males or non-pregnant females of 18 years of age, and in good general health, as determined by Investigator.
* Have 16 natural, gradable teeth and good dental health, as determined by Investigator.
* Have > 25% sites with GI scores > 2.
* Have average PI score > 2.
* Use of effective method of contraception for the duration of the study or permanently sterilized.
* Able and willing to comply with study requirements including following instructions on study treatment (drug) and returning for follow-up visits as required by the protocol.

Have full understanding of all elements of, and signature and dating of the written informed consent prior to the initiation of protocol specified procedures. Females with childbearing potential must have a negative pregnancy test before and during the study period. Sexually active females must be using an effective form of birth control. These methods include oral contraceptives ("the pill"), an intrauterine device (IUD), levonogestrol implants (Norplant®), medroxyprogesterone acetate injections (Depo-provera®) or contraceptive foam with a condom.

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria are not eligible for participation in this study:

* History, or current evidence, of any significant acute or chronic medical or psychiatric condition that, in the opinion of the Investigator, would render examination difficult or invalid or prevent the subject from active study participation.
* Treatment with antibiotic within the one (1) month period prior to the screening examination.
* Presence of heart murmur, history of rheumatic fever, valvular disease or prosthetic implant requiring antibiotic premedication.
* History of thyroid disease.
* Known sensitivity or allergy to iodine.
* Known sensitivity or allergy to shellfish.
* History of diabetes.
* History of autoimmune disease.
* Gross oral pathology (periodontal disease, rampant caries, tissue damage created by poor oral care or treatment, soft or hard tissue tumors) that, in the opinion of the Investigator, could influence the outcome of the study.
* Current signs or symptoms of mucosal tissue ulcerations or inflammation, or canker sores.
* Presence of orthodontic appliances or any removable appliance that impinges on the oral tissues being assessed.
* History of early onset periodontal disease or acute necrotizing ulcerative gingivitis.
* History of or current alcohol abuse that, in the opinion of the Investigator, could influence the outcome of the study.
* History of, or current drug abuse.
* Use of concomitant medication that, in the opinion of the Investigator, might interfere with the outcome of the study (e.g. antibiotics, immuno-suppressants, steroids, or therapeutic doses of non-steroidal anti-inflammatory agents, phenytoin, calcium antagonists, cyclosporine or coumadin).
* Concomitant therapy with another investigational drug or device without prior approval from the Sponsor within four (4) weeks prior to Visit 2 (Study Day 1).
* Concomitant endodontic or periodontal therapy other than prophylaxis in the past six (6) months.
* Females with childbearing potential with a positive pregnancy test, pregnant or nursing mothers, suspected pregnancy, or intention to become pregnant during the study.
* Unable and unwilling to comply with the informed consent process, to meet study requirements including following instructions on study treatment (drug), and to return for follow-up visits as required by the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14
Dates: Start 2006-10; Study Completion 2007-01

PRIMARY OUTCOMES:
Reduction of the Gingival Index values over a 12 weeks period.

SECONDARY OUTCOMES:
Reduction of the Plaque Index values over a 12 weeks period.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Friesen, DDS, Principal Investigator — University of Missouri at Kansas City, School of Dentistry
Locations (1):
- University of Missouri at Kansas City, School of Dentistry, Kansas City, Missouri, United States

REFERENCES:
- [Background] Guidance for Industry Gingivitis: Development and Evaluation of Drugs for Treatment or Prevention